CLINICAL TRIAL: NCT04257877
Title: Targeted Proteomic Analysis in the Plasma of Children With Diabetes Type 1 and Its Association With Peripheral Diabetic Neuropathy
Brief Title: Proteomic Analysis in Paediatric Diabetes Type 1 (PAPD)
Acronym: PAPD
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, Professor, Aristotle University Of Thessaloniki
Other Study IDs: 1.109/21.11.2018
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Type 1; Proteomics; Diabetic Peripheral Neuropathy
Keywords: plasma proteomics; children; diabetes type 1; nerve conduction
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Proteomics in plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes type 1: Patients= diabetes type1
  Interventions: Procedure: Blood sampling
- Healthy participants: Healthy participants = Control group
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood samples for proteomic analysis in plasma of both groups

SUMMARY:
The aim of the present study is to investigate a targeted proteomic analysis in plasma of children - of Greek origin- with type 1 diabetes (DT1) and its correlation with the electrophysiological findings that accompany diabetic peripheral neuropathy.

Diabetic neuropathy is the most frequent chronic complication in adults with DT1 and rarely appears in childhood. Nevertheless, cases of acute mononeuritis have been described at the time of diagnosis of DT1. According to recent reports several biomarkers, including proteomic analysis, have been proposed for the early detection of peripheral neuropathy in children and young adults with T1DM.

In the present study the researchers will attempt to investigate the role of biomarkers with targeted proteomic analysis in the plasma of children with DT1 in combination with an electrophysiological study, which includes a nerve conduction study, to detect early diabetic peripheral neuropathy, before the appearance of clinical manifestations.

ELIGIBILITY:
Inclusion Criteria:

1. Children with confirmed DT1 under insulin substitution therapy
2. Age 5-10 years
3. Good glycemic control with HbA1c ≤ 7.0%
4. Prepubertal patients
5. Absence of other diseases
6. Signed informed consent of the parents or guardians of patients

Exclusion Criteria:

1. Presence of organic cause for neuropathy
2. Presence of other chronic disease
3. Poor glycemic control

3. Medication

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Diabetes type 1 group
  * Good glycemic control with HbA1c ≤ 7.0%
  * Prepubertal patients (stage Tanner I :
  Estradiol E2 < 15pg/dl for girls, Testosterone T < 10ng/dl for boys)
  Healthy participants group:
  * Age 5-10 years
  * No medication
  * No acute or chronic disease
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Targeted proteomic analysis in children with DT1 (levels of certain plasma proteomics such as sorbitol, fructose, myo-inositol, scyllo-inositol, serine, lysine, tertadecanoic, palmitic, stearic, eicosanoic fatty acids) | 2018-2020

SECONDARY OUTCOMES:
Electrophysiological study | 2018-2020
  electrophysiological findings such as nerve conduction velocity indicative of peripheral neuropathy.
  - Correlation of proteomic analysis results with electrophysiological findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Pediatric Endocrinology, Diabetes and Metabolism-2nd Department of Pediatrics, School of Medicine, Faculty of Health Sciences, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donaghue KC, Bonney M, Simpson JM, Schwingshandl J, Fung AT, Howard NJ, Silink M. Autonomic and peripheral nerve function in adolescents with and without diabetes. Diabet Med. 1993 Aug-Sep;10(7):664-71. doi: 10.1111/j.1464-5491.1993.tb00142.x. PMID 8403830
- [Background] Donaghue KC, Silink M. Diabetic neuropathy in childhood. Diabetes Nutr Metab. 1999 Apr;12(2):154-60. No abstract available. PMID 10554898
- [Background] Otto-Buczkowska E, Kazibutowska Z, Soltyk J, Machnica L. Neuropathy and type 1 diabetes mellitus. Pediatr Endocrinol Diabetes Metab. 2008;14(2):109-16. PMID 18721498
- [Background] Said G, Bigo A, Ameri A, Gayno JP, Elgrably F, Chanson P, Slama G. Uncommon early-onset neuropathy in diabetic patients. J Neurol. 1998 Feb;245(2):61-8. doi: 10.1007/s004150050179. PMID 9507409
- [Background] Rangel MA, Baptista C, Santos F, Real MV, Campos RA, Leite AL. Acute mononeuropathy in a child with newly diagnosed type 1 diabetes mellitus. J Pediatr Endocrinol Metab. 2015 Mar;28(3-4):341-4. doi: 10.1515/jpem-2014-0049. PMID 25153576
- [Background] Louraki M, Karayianni C, Kanaka-Gantenbein C, Katsalouli M, Karavanaki K. Peripheral neuropathy in children with type 1 diabetes. Diabetes Metab. 2012 Oct;38(4):281-9. doi: 10.1016/j.diabet.2012.02.006. Epub 2012 Apr 12. PMID 22503144
- [Background] Albers JW, Herman WH, Pop-Busui R, Feldman EL, Martin CL, Cleary PA, Waberski BH, Lachin JM; Diabetes Control and Complications Trial /Epidemiology of Diabetes Interventions and Complications Research Group. Effect of prior intensive insulin treatment during the Diabetes Control and Complications Trial (DCCT) on peripheral neuropathy in type 1 diabetes during the Epidemiology of Diabetes Interventions and Complications (EDIC) Study. Diabetes Care. 2010 May;33(5):1090-6. doi: 10.2337/dc09-1941. Epub 2010 Feb 11. PMID 20150297
- [Background] Barkai L, Kempler P, Vamosi I, Lukacs K, Marton A, Keresztes K. Peripheral sensory nerve dysfunction in children and adolescents with type 1 diabetes mellitus. Diabet Med. 1998 Mar;15(3):228-33. doi: 10.1002/(SICI)1096-9136(199803)15:33.0.CO;2-8. PMID 9545124
- [Background] Sosenko JM, Boulton AJ, Kubrusly DB, Weintraub JK, Skyler JS. The vibratory perception threshold in young diabetic patients: associations with glycemia and puberty. Diabetes Care. 1985 Nov-Dec;8(6):605-7. doi: 10.2337/diacare.8.6.605. PMID 4075949
- [Background] Mayhew JA, Gillon KR, Hawthorne JN. Free and lipid inositol, sorbitol and sugars in sciatic nerve obtained post-mortem from diabetic patients and control subjects. Diabetologia. 1983 Jan;24(1):13-5. doi: 10.1007/BF00275940. PMID 6825977
- [Background] Mistry KP, Beyer-Mears A, Diecke FP. Mechanisms for D-glucose inhibition of myo-inositol influx into rat lens. Diabetes. 1993 Dec;42(12):1737-44. doi: 10.2337/diab.42.12.1737. PMID 8243820
- [Background] Brownlee M, Vlassara H, Cerami A. Nonenzymatic glycosylation products on collagen covalently trap low-density lipoprotein. Diabetes. 1985 Sep;34(9):938-41. doi: 10.2337/diab.34.9.938. PMID 4029512
- [Background] Nery Ferreira BE, Silva IN, de Oliveira JT. High prevalence of diabetic polyneuropathy in a group of Brazilian children with type 1 diabetes mellitus. J Pediatr Endocrinol Metab. 2005 Nov;18(11):1087-94. doi: 10.1515/jpem.2005.18.11.1087. PMID 16459455
- [Background] Lee SS, Han HS, Kim H. A 5-yr follow-up nerve conduction study for the detection of subclinical diabetic neuropathy in children with newly diagnosed insulin-dependent diabetes mellitus. Pediatr Diabetes. 2010 Dec;11(8):521-8. doi: 10.1111/j.1399-5448.2009.00636.x. Epub 2010 Aug 15. PMID 20723100
- [Background] Hyllienmark L, Alstrand N, Jonsson B, Ludvigsson J, Cooray G, Wahlberg-Topp J. Early electrophysiological abnormalities and clinical neuropathy: a prospective study in patients with type 1 diabetes. Diabetes Care. 2013 Oct;36(10):3187-94. doi: 10.2337/dc12-2226. Epub 2013 May 30. PMID 23723354
- [Background] Albers JW, Herman WH, Pop-Busui R, Martin CL, Cleary P, Waberski B; Diabetes Control and Complications Trial (DCCT)/Epidemiology of Diabetes Intervention and Complications (EDIC) Research Group. Subclinical neuropathy among Diabetes Control and Complications Trial participants without diagnosable neuropathy at trial completion: possible predictors of incident neuropathy? Diabetes Care. 2007 Oct;30(10):2613-8. doi: 10.2337/dc07-0850. Epub 2007 Jul 20. PMID 17644617
- [Background] Toopchizadeh V, Shiva S, Khiabani NY, Ghergherechi R. Electrophysiologic pattern and prevalence of subclinical peripheral neuropathy in children and adolescents with type I diabetes mellitus in Iran. Saudi Med J. 2016 Mar;37(3):299-303. doi: 10.15537/smj.2016.3.13625. PMID 26905353
- [Background] Hajas G, Kissova V, Tirpakova A. A 10-yr follow-up study for the detection of peripheral neuropathy in young patients with type 1 diabetes. Pediatr Diabetes. 2016 Dec;17(8):632-641. doi: 10.1111/pedi.12382. Epub 2016 Mar 29. PMID 27028140
- [Background] Giannopoulou EG, Garbis SD, Vlahou A, Kossida S, Lepouras G, Manolakos ES. Proteomic feature maps: a new visualization approach in proteomics analysis. J Biomed Inform. 2009 Aug;42(4):644-53. doi: 10.1016/j.jbi.2009.01.007. Epub 2009 Feb 4. PMID 19535004
- [Background] Balderas C, Ruperez FJ, Ibanez E, Senorans J, Guerrero-Fernandez J, Casado IG, Gracia-Bouthelier R, Garcia A, Barbas C. Plasma and urine metabolic fingerprinting of type 1 diabetic children. Electrophoresis. 2013 Oct;34(19):2882-90. doi: 10.1002/elps.201300062. Epub 2013 Sep 10. PMID 23857511
- [Background] Bain JR, Stevens RD, Wenner BR, Ilkayeva O, Muoio DM, Newgard CB. Metabolomics applied to diabetes research: moving from information to knowledge. Diabetes. 2009 Nov;58(11):2429-43. doi: 10.2337/db09-0580. No abstract available. PMID 19875619
- [Background] Wallaschofski H. What will metabolomics studies mean to endocrinology? J Endocrinol. 2012 Oct;215(1):1-2. doi: 10.1530/JOE-12-0270. Epub 2012 Jul 3. No abstract available. PMID 22761276
- [Background] Suhre K, Meisinger C, Doring A, Altmaier E, Belcredi P, Gieger C, Chang D, Milburn MV, Gall WE, Weinberger KM, Mewes HW, Hrabe de Angelis M, Wichmann HE, Kronenberg F, Adamski J, Illig T. Metabolic footprint of diabetes: a multiplatform metabolomics study in an epidemiological setting. PLoS One. 2010 Nov 11;5(11):e13953. doi: 10.1371/journal.pone.0013953. PMID 21085649
- [Background] McKillop AM, Flatt PR. Emerging applications of metabolomic and genomic profiling in diabetic clinical medicine. Diabetes Care. 2011 Dec;34(12):2624-30. doi: 10.2337/dc11-0837. PMID 22110171
- [Background] Lanza IR, Zhang S, Ward LE, Karakelides H, Raftery D, Nair KS. Quantitative metabolomics by H-NMR and LC-MS/MS confirms altered metabolic pathways in diabetes. PLoS One. 2010 May 10;5(5):e10538. doi: 10.1371/journal.pone.0010538. PMID 20479934
- [Background] van der Kloet FM, Bobeldijk I, Verheij ER, Jellema RH. Analytical error reduction using single point calibration for accurate and precise metabolomic phenotyping. J Proteome Res. 2009 Nov;8(11):5132-41. doi: 10.1021/pr900499r. PMID 19754161
- [Background] Dutta T, Chai HS, Ward LE, Ghosh A, Persson XM, Ford GC, Kudva YC, Sun Z, Asmann YW, Kocher JP, Nair KS. Concordance of changes in metabolic pathways based on plasma metabolomics and skeletal muscle transcriptomics in type 1 diabetes. Diabetes. 2012 May;61(5):1004-16. doi: 10.2337/db11-0874. Epub 2012 Mar 13. PMID 22415876
- [Background] Zhang S, Zheng C, Lanza IR, Nair KS, Raftery D, Vitek O. Interdependence of signal processing and analysis of urine 1H NMR spectra for metabolic profiling. Anal Chem. 2009 Aug 1;81(15):6080-8. doi: 10.1021/ac900424c. PMID 19950923
- [Background] Zhang S, Nagana Gowda GA, Asiago V, Shanaiah N, Barbas C, Raftery D. Correlative and quantitative 1H NMR-based metabolomics reveals specific metabolic pathway disturbances in diabetic rats. Anal Biochem. 2008 Dec 1;383(1):76-84. doi: 10.1016/j.ab.2008.07.041. Epub 2008 Aug 20. PMID 18775407
- [Background] Moraes EP, Ruperez FJ, Plaza M, Herrero M, Barbas C. Metabolomic assessment with CE-MS of the nutraceutical effect of Cystoseira spp extracts in an animal model. Electrophoresis. 2011 Aug;32(15):2055-62. doi: 10.1002/elps.201000546. PMID 21792987
- [Background] Godzien J, Ciborowski M, Angulo S, Ruperez FJ, Martinez MP, Senorans FJ, Cifuentes A, Ibanez E, Barbas C. Metabolomic approach with LC-QTOF to study the effect of a nutraceutical treatment on urine of diabetic rats. J Proteome Res. 2011 Feb 4;10(2):837-44. doi: 10.1021/pr100993x. Epub 2010 Dec 20. PMID 21087057
- [Background] Balderas C, Villasenor A, Garcia A, Ruperez FJ, Ibanez E, Senorans J, Guerrero-Fernandez J, Gonzalez-Casado I, Gracia-Bouthelier R, Barbas C. Metabolomic approach to the nutraceutical effect of rosemary extract plus Omega-3 PUFAs in diabetic children with capillary electrophoresis. J Pharm Biomed Anal. 2010 Dec 15;53(5):1298-304. doi: 10.1016/j.jpba.2010.07.034. Epub 2010 Jul 30. PMID 20719450
- [Background] Vallejo M, Angulo S, Garcia-Martinez D, Garcia A, Barbas C. New perspective of diabetes response to an antioxidant treatment through metabolic fingerprinting of urine by capillary electrophoresis. J Chromatogr A. 2008 Apr 11;1187(1-2):267-74. doi: 10.1016/j.chroma.2008.02.024. Epub 2008 Feb 12. PMID 18316089
- [Background] Bervoets L, Massa G, Guedens W, Louis E, Noben JP, Adriaensens P. Metabolic profiling of type 1 diabetes mellitus in children and adolescents: a case-control study. Diabetol Metab Syndr. 2017 Jun 26;9:48. doi: 10.1186/s13098-017-0246-9. eCollection 2017. PMID 28674557
- [Background] Biessels GJ, Bril V, Calcutt NA, Cameron NE, Cotter MA, Dobrowsky R, Feldman EL, Fernyhough P, Jakobsen J, Malik RA, Mizisin AP, Oates PJ, Obrosova IG, Pop-Busui R, Russell JW, Sima AA, Stevens MJ, Schmidt RE, Tesfaye S, Veves A, Vinik AI, Wright DE, Yagihashi S, Yorek MA, Ziegler D, Zochodne DW. Phenotyping animal models of diabetic neuropathy: a consensus statement of the diabetic neuropathy study group of the EASD (Neurodiab). J Peripher Nerv Syst. 2014 Jun;19(2):77-87. doi: 10.1111/jns5.12072. PMID 24934510
- [Background] Zhang L, Yu C, Vasquez FE, Galeva N, Onyango I, Swerdlow RH, Dobrowsky RT. Hyperglycemia alters the schwann cell mitochondrial proteome and decreases coupled respiration in the absence of superoxide production. J Proteome Res. 2010 Jan;9(1):458-71. doi: 10.1021/pr900818g. PMID 19905032
- See also: Spiros Garbis, Associate Professor , Head of Proteomics Unit for Cancer Sciences, Centre for Proteomics Research, Institute for Life Sciences, UK — https://www.southampton.ac.uk/medicine/research/staff/sdg2e11.page